CLINICAL TRIAL: NCT05429892
Title: FRESH Delivers: An Innovative Approach to Reducing Tobacco Use Among Rural Smokers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 273441
Record Dates: First submitted 2022-05-23; First posted 2022-06-23 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Tobacco Cessation; Tobacco Dependence; Food Security
Keywords: food security; smoking cessation; social change; motivational counseling; home food delivery; tobacco biomarkers
MeSH Terms: conditions — Tobacco Use Cessation; Tobacco Use Disorder; Smoking Cessation

STUDY DESIGN:
Intervention Model Description: The 3-arm trial (180 smokers per arm) will enroll 540 smokers in Chicot, Desha, Lee, and Phillips and deliver the intervention over 6 months. The study is powered to examine our primary outcome, cotinine-verified 7-day point prevalence abstinence, after 6 months and we will conduct a 12-month follow-up survey. The secondary outcome will be food security. 180 smokers aged 21-75 will be randomized to each condition.
Who Masked: Participant, Care Provider
Masking Description: The community health workers who will deliver the intervention will not have access to the randomization information. The participants will also not have access to the information the randomization information.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TRTsocialmot1 arm (Experimental): Smokers will receive real-time video-based motivational counseling and home-based food delivery or grocery store gift card.
  Participants will receive educational material.
  Interventions: Behavioral: Smoking cessation counseling and food delivery
- TRTmot3 arm (Active Comparator): Smokers will receive real-time video-based motivational counseling only.
  Participants will receive educational material.
  Interventions: Behavioral: Smoking cessation counseling
- TRTsocial2 arm (Active Comparator): Smokers will receive home-based food delivery only or grocery store gift card.
  Participants will receive educational material.
  Interventions: Behavioral: Food delivery

INTERVENTIONS:
Behavioral: Smoking cessation counseling and food delivery — The community health workers will delivery three 30-minute sessions during intervention months 1 through 6 (1,3,6 months) to provide interpersonal level support for smoking cessation. The community health workers will conduct real-time video motivational counseling to clients. The community health workers will implement the 5As (Ask, Advise, Assess, Assist, Arrange) and support smokers in quitting, if ready, and build confidence toward quitting if they are uncertain about change.
  Smokers enrolled in the TRTsocialmot1 arm will be provided with food boxes or grocery store gift card at 1,3, and 6 months. Healthy meal preparation instructions will be included and delivery by project staff and will reduce transportation barriers to food access rural counties.
  Participants will receive educational materials at 1, 3, and 6 months.
  Other Names: TRTsocialmot1
  Arms: TRTsocialmot1 arm
Behavioral: Smoking cessation counseling — The community health workers will deliver three 30-minute sessions during intervention months 1 through 6 (1,3,6 months) to provide interpersonal level support for smoking cessation. The community health workers will conduct real-time video motivational counseling to clients. The community health workers will implement the 5As (Ask, Advise, Assess, Assist, Arrange) and support smokers in quitting, if ready, and build confidence toward quitting if they are uncertain about change.
  Participants will receive educational materials at 1, 3, and 6 months.
  Other Names: TRTmot3 arm
  Arms: TRTmot3 arm
Behavioral: Food delivery — Smokers enrolled in the TRTsocial2 arm will be provided with food boxes or grocery store gift card at 1, 3, and 6 months Healthy meal preparation instructions will be included and delivery by project staff and will reduce transportation barriers to food access rural counties.
  Participants will receive educational materials.
  Other Names: TRTsocial2
  Arms: TRTsocial2 arm

SUMMARY:
The long-term goal of FRESH Delivers is to fill a critical gap in knowledge on the role of a home-based food delivery social intervention in the elimination of tobacco-caused cancer health burdens. The central hypothesis is that smokers who receive real-time video-based motivational counseling and home-based food deliveries will have greater cotinine-verified 7-day point prevalence abstinence than those who receive real-time video-based motivational counseling alone or home food delivery alone. The rationale for this approach is that studies show increased odds of smoking cessation with increasing food security.

DETAILED DESCRIPTION:
The central hypothesis is that smokers who receive real-time video-based motivational counseling and home-based food deliveries will have greater cotinine-verified 7-day point prevalence abstinence than those who receive real-time video-based motivational counseling alone or home food delivery alone. The rationale for this approach is that studies show increased odds of smoking cessation with increasing food security. Prior studies have largely ignored intervening on social conditions that perpetuate chronic disease burdens, resulting in repeated failures to reach smokers in low-resource counties with effective interventions that help them quit smoking. A limited number of interventions that aimed to increase food security also resulted in increased fruit and vegetable consumption and decreased body mass index. But, none have examined the effects of providing food security as a means to help smokers quit. The aims are:

Aim 1. Test the efficacy of a social change intervention (home food delivery) on smoking abstinence using a 3-arm randomized controlled design. H1.1: Smokers who receive real-time video-based motivational counseling and home-based food delivery will have greater cotinine-verified 7-day point prevalence abstinence than smokers who receive real-time video-based motivational counseling alone or home food delivery alone.

Aim 2. Examine changes in measures of cigarette abuse liability across treatment groups. H2.1: Smokers in the real-time video-based motivational counseling and home-based food delivery intervention will have: 1) fewer signs of nicotine dependence, cravings, and withdrawal and lower levels of biomarkers of tobacco exposure (carbon monoxide, cotinine, trans-3'-hydroxycotinine) and tobacco harm (acrolein, acetaldehyde, benzaldehyde, and formaldehyde) than smokers who receive real-time video-based motivational counseling alone or home food delivery alone. H2.2: Smokers with higher social stressors will show greater signs of nicotine dependence, cravings, and withdrawal and higher levels of biomarkers of tobacco exposure and harm.

Aim 3. Examine the extent to which a home food delivery intervention improves recruitment and retention of smokers in the treatment condition. H3.1: Smokers in the real-time video-based motivational counseling and home-based food delivery intervention will have greater reach, dose, and successful referrals compared to smokers who receive motivational counseling alone or home food delivery alone.

Impact. The novel home-based food delivery with real-time video-based motivational counseling intervention could increase access to cessation interventions in rural counties where interventions are lacking and encourage Americans to participate in interventions that meets a basic need, food security, thus improving social conditions, increasing smoking cessation, and potentially eliminating the risk for cancer health burdens.

ELIGIBILITY:
Inclusion Criteria:

* Currently smoke regularly for at least 1 year with a verified carbon monoxide level of 5 ppm or greater
* Live in Desha, Phillips, Chicot, or Lee Counties
* Aged 21 to 75
* Speak English
* Interest in quitting
* Provide written/online informed consent
* Working phone, home address, and email
* Willingness to use a study provided tablet/phone service
* Willingness to report COVID-19 symptoms as appropriate to assure everyone's safety during a personal visit.

Exclusion Criteria:

• Persons who do not meet the above criteria.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 540 (Estimated)
Dates: Start 2023-08-09 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Cotinine verified- 7 day point prevalence abstinence | Changes from baseline cigarette prevalence at 6 months
  The study is powered to examine changes in our primary outcome, cotinine-verified 7-day point prevalence abstinence using survey data and collecting a saliva sample.

SECONDARY OUTCOMES:
Food security | Changes from baseline food security at 6 months
  The secondary outcome will be food security measured using the US household food security 6-item survey. Scores of 0-1= high to marginal food security; 2-4= low food security; 5-6= very low food security.

OTHER OUTCOMES:
Abuse liability - nicotine dependence | Changes from baseline nicotine dependence at 6 months
  Examine changes in measures of cigarette abuse liability across treatment groups. Abuse liability will be measured using a 6-item nicotine dependence (Fagerstrom Test for Nicotine Dependence) scale on surveys. Scores of 8-10=very high dependence; 6-7= high ; 5= moderate; 3-4= low; 0-2= very low dependence.
Abuse liability - carbon monoxide | Changes from baseline carbon monoxide at 6 months
  Examine changes in measures of cigarette abuse liability across treatment groups. Abuse liability will be measured using carbon monoxide measured via the Smokerlyzer® monitors. Higher carbon monoxide scores mean greater exposure to tobacco.
Abuse liability - cotinine | Changes from baseline cotinine at 6 months
  Examine changes in measures of cigarette abuse liability across treatment groups. Abuse liability will be measured by collecting saliva that will allow us to assess cotinine levels. Higher cotinine levels mean greater exposure tobacco.
Abuse liability - trans-3'-hydroxycotinine | Changes from baseline trans-3'-hydroxycotinine at 6 months
  Examine changes in measures of cigarette abuse liability across treatment groups. Abuse liability will be measured by collecting saliva that will allow us to assess - trans-3'-hydroxycotinine levels. Higher levels mean greater exposure to tobacco.
Abuse liability - cravings | Changes from baseline cravings at 6 months
  Examine changes in measures of cigarette abuse liability across treatment groups. Abuse liability will be measured using the 10-item brief questionnaire of smoking urges. Scores range from 1 (strongly disagree) to 7 (strongly agree) ad result in two factors related to specific items in the scale. The higher the score, the stronger to urge.
Abuse liability - withdrawal | Changes from baseline withdrawal at 6 months
  Examine changes in measures of cigarette abuse liability across treatment groups. Abuse liability will be measured using the 6-item Minnesota withdrawal scale (2021). Scores range from 0=none to 4=severe. The higher the score the more severe the withdrawal.
Abuse liability - acrolein | Changes from baseline acrolein at 6 months
  Examine changes in measures of cigarette abuse liability across treatment groups. Abuse liability will be measured by collecting saliva that will allow us to assess -acrolein levels. Higher levels mean greater exposure to this tobacco toxin.
Abuse liability - benzaldehyde | Changes from baseline benzaldehyde at 6 months
  Examine changes in measures of cigarette abuse liability across treatment groups. Abuse liability will be measured by collection saliva that will allow us to assess benzaldehyde levels. Higher levels mean greater exposure to this tobacco toxin.
Abuse liability - formaldehyde | Changes from baseline formaldehyde at 6 months
  Examine changes in measures of cigarette abuse liability across treatment groups. Abuse liability will be measured by collection saliva that will allow us to assess formaldehyde levels. Higher levels mean greater exposure to this tobacco toxin.
Recruitment and retention- reach | Monthly until study completion, on average 1 year.
  Examine reach to participants. Reach will be assessed by calculating # participants enrolled in the study each month. Staff will review completed consent forms and baseline surveys monthly.
Recruitment and retention-dose delivered | Monthly until study completion, on average 1 year.
  Examine dose of the intervention delivered to participants. Dose delivered will be assessed by calculating the number of intervention activities delivered (motivational counseling, food delivery). Staff will complete a process tracking form after the delivery of each intervention activity.
Recruitment and retention-dose received | At 6 months.
  Examine dose of the intervention received by participants. Dose received will be assessed by calculating the participant report of number of interventions received (motivational counseling, food delivery). Participants will be asked about the interventions received on the 6-month survey.
Recruitment and retention- successful referral | Monthly until study completion, on average 1 year.
  Examine successful referral of participants to the study. Staff will document the number of persons who enrolled in the study who were referred by an enrolled study participant.

CONTACTS AND LOCATIONS:
Overall Officials: Pebbles Fagan, PhD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: Yes
We will coordinate these efforts with the NIMHD research coordinating center to determine what data will be shared across studies.
Supporting Information: Study Protocol
Time Frame: At the end of the study
Access Criteria: Contact the PI for the protocol and obtain instructions on how to access. Persons must complete registration.